CLINICAL TRIAL: NCT05934929
Title: Contribution of Residual Tumour DNA Testing on the Surgical Bed of Squamous Cell Carcinomas of the Oral Cavity
Brief Title: Contribution of Residual Tumour DNA Testing on the Surgical Bed
Acronym: MARGINS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Henri Becquerel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHB23.01; 2023-A00567-38 (Other: ANSM)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
Keywords: oral cavity; squamous cell carcinoma; residual tumor DNA; head and neck surgery
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- circulating tumor DNA detection on operating bed (Experimental): biological assessment on operating bed to detect residual circulating tumor DNA
  Interventions: Other: Circulating tumor DNA detection

INTERVENTIONS:
Other: Circulating tumor DNA detection — biological assessment on operating bed to detect residual circulating tumor DNA

SUMMARY:
The aim of this study is to evaluate the interest of residual tumour DNA research in the operating bed after squamous cell carcinoma excision.

DETAILED DESCRIPTION:
Squamous cell carcinomas of the oral cavity have a poor prognosis. The 5-year loco-regional recurrence rate is 45%. Surgery remains the standard treatment. The presence of invasive or insufficient surgical margins is an important histopronostic factor.

Current tools for intraoperative detection of insufficient margins have a very low sensitivity of around 10%. The aim here is to develop a more sensitive tool by looking for the presence of residual tumour DNA in the entire operating bed after squamous cell carcinoma excision

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient with T1 to T4 squamous cell carcinoma of the oral cavity, regardless of lymph node status (all N) M0, operable
* 18 years of age or older
* Member or beneficiary of a social security scheme.

Exclusion Criteria:

* Absence of signed informed consent
* Patient of protected age
* Psychosocial problems
* Not affiliated to or benefiting from a social security scheme
* Previous cervical irradiation
* Pregnant or breast-feeding women
* Patient unable to understand the study for any reason or to comply with the constraints of the trial (language, psychological, geographical problems, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2027-12-29 (Estimated)

PRIMARY OUTCOMES:
Residual tumro DNA on operating bed | during the surgery
  Proportion of patients with residual tumour DNA on the operating bed according to the presence or absence of adverse histological factors

SECONDARY OUTCOMES:
Survival without locoregional recurrence rate | 24 months
  Proportion of patients with circulating tumour DNA and in the cervical lymphatic drainage fluid or circulating blood according to the presence or absence of residual tumour DNA on the operating bed

CONTACTS AND LOCATIONS:
Overall Officials: Lise-Marie Roussel, MD, Principal Investigator — Centre Henri Becquerel
Locations (2):
- France (2):
  - CHU Rouen, Rouen
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No